CLINICAL TRIAL: NCT04732351
Title: Observational Multicenter Registry to Assess the Enefits of Active Sentry Handpiece During Cataract Surgery With the Centurion Phacoemulsifier (SASCA)
Brief Title: Evaluation of the Active Sentry System During Cataract Surgery With the Centurion Phacoemulsifier
Acronym: SASCA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201099; 57203277 (Other Grant/Funding Number: Alcon EMA IIT)
Record Dates: First submitted 2021-01-29; First posted 2021-02-01 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cataract Surgery
Keywords: Cataract surgery; phacoemulsification; Cumulated dissipated energy; Active Sentry; Centurion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active sentry: Cataract procedures conducted with the active Sentry handpiece
- Non-active sentry: Cataract procedures conducted with an handpiece different from the Active Sentry Handpiece

SUMMARY:
Each new generation of phacoemulsification system has aimed to optimize the control of fluidics and the delivery of energy during phacoemulsification. Nicoli CM et al., (J Cataract Refract Surg 2016;42:157-162) suggested a better anterior chamber stability when using an active fluidics system. Malik PK et al., (Eye and Vision 2017;4:22) showed that using an IOP based phacoemulsification system in association with the use of an Intrepid balanced tip provides a reduction in CDE (Cumulated Dissipated Energy and EFU (Estimated Fluid Usage). It has also been shown that a lower CDE provides obvious benefits: less endothelium cells damages and lower complication rates (Mady MA et al., Clin.Ophthalmol. 2012; 6:503-10).

The latest technologies, i.e. the Active Sentry Handpiece and Hybrid tips, have been introduced to further improve the safety of phacoemulsification. The Active Sentry system has moved pressure sensors closer to the operated eye, hence further reducing the risk of surge during procedures. (Thorne A et al. Phacoemulsifier occlusion break surge volume reduction, J Cataract Refract Surg. 2018;44:1491-1496). The Hybrid tips have been designed to prevent posterior capsule rupture in the event of contact with the capsule.

This new technology allows phacoemulsification procedures under reduced infusion pressures and a "high-vacuum - low energy" strategy which may lead to a safer procedure.

Data from this study will try to demonstrate that cataract surgeries with Active Sentry will need less CDE and therefore may be safer, due to the surge effects decrease. This CDE parameter will be analysed according to differents subgroups: Presence of hybrid tip or balanced tip, cataract score based on the WHO nuclear grading recommendation (Thylefors B et al., (2002) The WHO Cataract Grading Group, Ophthalmic Epidemiology, 9:2, 83-95) The recent experiences conducted in real world condition in different sites have suggested that Centurion with AS was able to improved settings: maximum vacuum and UltraSound (US) time reduction and as a consequence a 20 to 30% CDE reduction.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients undergoing unilateral or bilateral cataract surgery with the Centurion phacoemulsifier, with the ability to give informed consent.
* Patients will undergo the cataract surgery with or without the Active Sentry module and with or without hybrid tip according to centers practice.
* Patients will undergo a cataract scoring (nuclear grade 1 to 3) prior surgery as described in the WHO recommendation:

Exclusion Criteria:

* Patients with :
* pupil dilation <5mm
* zonular defects
* corneal opacities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo a cataract surgery in routine
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Mean CDE (Cumulated Dissipated Energy) | The day of the cataract procedure
  Mean CDE measured by the phacoemulsifier in different groups according to baseline patients and/or eyes characteristics (nuclear cataract grading etc...)

SECONDARY OUTCOMES:
Mean total procedure duration | The day of the cataract procedure
  Mean total duration of each procedure in different groups
Mean total Ultrasound time (US time) | The day of the procedure
  Mean total Ultrasound time (US time) in different groups
Mean procedure settings | The day of the procedure
  Mean procedure settings : infusion pressure, aspiration flow and vacuum levels
Mean BSS volume | The day of the procedure
Frequency of adverse events | The day of the procedure
  Mean frequency of adverse events during procedures, including posterior capsule ruptures

CONTACTS AND LOCATIONS:
Overall Officials: Antoine BREZIN, PhD & MD, Principal Investigator — Hopital Cochin, Ophthalmology, Paris
Locations (1):
- Ophtalmopôle, Hôpital Cochin, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brezin AP, Monnet D, Lignereux F, Rozot P, Jilet L, Abdoul H. Impact of a handpiece with a built-in fluidics pressure sensor on phacoemulsification: a multicentre prospective comparative study. BMJ Open Ophthalmol. 2023 Nov;8(1):e001431. doi: 10.1136/bmjophth-2023-001431. PMID 37973548